CLINICAL TRIAL: NCT03098407
Title: A Pilot Randomized Comparative Effectiveness Clinical Trial of Buprenorphine vs. Methadone for the Treatment of Opioid Dependence in Pregnancy.
Brief Title: Opioid Dependence Treatment Therapies in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Krans, MD, Assistant Professor, Department of Obstetrics, Gynecology & Reproductive Sciences, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO16020403; 1K23DA038789-01A1 (NIH)
Record Dates: First submitted 2016-10-24; First posted 2017-03-31 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Opioid-Related Disorders; Pregnancy
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Methadone

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buprenorphine Maintenance Treatment (Other): Buprenorphine Maintenance Treatment patients will receive instructions regarding a follow-up, outpatient appointment with the Pregnancy Recovery Center at Magee-Womens Hospital, which specializes in Opioid maintenance treatment for pregnant patients, for the next day following enrollment in the study for induction onto buprenorphine maintenance treatment.
  Interventions: Drug: Buprenorphine
- Methadone Maintenance Treatment (Other): Methadone Maintenance Treatment patients will be immediately admitted to Magee-Womens Hospital for an inpatient induction onto methadone maintenance treatment.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Buprenorphine — This is a pilot study to establish the feasibility and acceptability of a randomized comparative effectiveness clinical trial comparing office-based buprenorphine vs. federally licensed methadone treatment programs for OD pregnant women.
  Arms: Buprenorphine Maintenance Treatment
Drug: Methadone — This is a pilot study to establish the feasibility and acceptability of a randomized comparative effectiveness clinical trial comparing office-based buprenorphine vs. federally licensed methadone treatment programs for OD pregnant women.
  Arms: Methadone Maintenance Treatment

SUMMARY:
The incidence of opioid dependence in pregnancy increased over the last decade from 1.2 to 5.8 per 1,000 hospital births per year.1 While methadone is the current, standard treatment for opioid dependent (OD) pregnant women, buprenorphine recently emerged as an alternative. In a recent clinical trial (MOTHER), buprenorphine was associated with superior neonatal outcomes such as shorter duration of treatment for neonatal abstinence syndrome (NAS) compared to methadone. However, buprenorphine was also associated with greater study discontinuation (33% vs. 18%) and illicit opioid use (33% vs. 23%) compared to methadone. Treatment dropout often leads to relapse and resumption of high-risk behaviors, overshadowing any short-term improvement in neonatal outcomes. Therefore, The goal of this K23 proposal is to conduct a pilot study to establish the feasibility and acceptability of a randomized comparative effectiveness clinical trial comparing office-based buprenorphine vs. federally licensed methadone programs for the treatment of OD pregnant women.

A pilot study is critical to develop the outcome measures, assessment tools and participant tracking techniques necessary for a future, large-scale comparative effectiveness clinical trial. An examination of feasibility and acceptability will also allow use to characterize the subpopulations of OD pregnant women willing to participate in treatment randomization, identify patient and provider characteristics associated with established treatment preferences and inform the development of strategies to improve participation and enhance the generalizability of the future large-scale clinical trial.

DETAILED DESCRIPTION:
Objective:

The goal of this proposal is to conduct a pilot study to establish the feasibility and acceptability of a randomized comparative effectiveness clinical trial comparing office-based buprenorphine vs. federally licensed methadone programs for the treatment of opioid dependent pregnant women.

Specific Aims:

Aim 1: Evaluate the feasibility of conducting a randomized study comparing office-based buprenorphine vs. federally licensed methadone programs for the treatment of OD pregnant women. OD pregnant women (n=50) will be randomized (1:1) to office-based buprenorphine vs. a federally licensed methadone program. Feasibility will be assessed by measuring the proportion of OD pregnant women who are eligible, who enroll, who remain in the study and by the ability to monitor treatment program factors (e.g. compliance with treatment provider/facility visits, counseling sessions, prenatal care visits, social services involvement) and maternal treatment outcomes such as treatment retention, illicit drug use and HIV risk behavior.

Aim 2: Describe the perspectives of OD pregnant women and their providers regarding buprenorphine vs. methadone for the treatment of opioid dependence in pregnancy. Study acceptability will be assessed by conducting qualitative semi-structured interviews with three groups: (1) pilot participants to determine their satisfaction with the assigned treatment program and identify mismatches between treatment program services and participants' needs; (2) prenatal care and opioid treatment providers to identify ways to improve the treatment process in pregnancy and to suggest ideas for care coordination; (3) OD pregnant women who are ineligible or who choose not to participate in the pilot trial will also be asked to participate in an interview to gain a broader perspective of attitudes and perspectives regarding opioid treatment programs in pregnancy.

Aim 3: Identify barriers and facilitators to treatment retention in the postpartum period and identify key functional outcomes relevant to reductions in illicit drug use during pregnancy. Illicit drug use relapse is most common in the immediate postpartum period when stresses associated with motherhood are the greatest. Therefore, pilot participants will be followed at 3, 6, 9 and 12 weeks postpartum to identify barriers and facilitators specific to the postpartum period that may impact treatment retention. The relationship between postpartum treatment retention and maternal functional outcomes will also be explored (e.g. breastfeeding, postpartum depression, motherhood satisfaction, infant custody, employment, and criminality).

Background:

The incidence of opioid dependence in pregnancy increased over the last decade from 1.2 to 5.8 per 1,000 hospital births per year. While methadone is the current, standard treatment for opioid dependent (OD) pregnant women, buprenorphine recently emerged as an alternative. In a recent clinical trial (MOTHER), buprenorphine was associated with superior neonatal outcomes such as shorter duration of treatment for neonatal abstinence syndrome (NAS) compared to methadone. However, buprenorphine was also associated with greater study discontinuation (33% vs. 18%) and illicit opioid use (33% vs. 23%) compared to methadone. Treatment dropout often leads to relapse and resumption of high-risk behaviors, overshadowing any short-term improvement in neonatal outcomes. Therefore, the next research question that emerges is which is the most effective treatment (buprenorphine vs. methadone) for a particular patient during pregnancy?

In clinical settings, differences in maternal characteristics, treatment program structure and patient and provider preferences may surpass the impact of pharmacology on maternal treatment outcomes (treatment retention, illicit drug use, HIV risk behavior). Buprenorphine is dispensed in office-based settings by a variety of providers and with less regulatory oversight than methadone. Methadone is dispensed from federally licensed facilities that often incorporate counseling and support services into treatment protocols. Successful office-based treatment relies on shared power and responsibility, close patient-provider relationships and careful attention to psychosocial co-morbidities. Failure to match patient problem severity to differences in treatment program structure may contribute to adverse maternal outcomes. Therefore, to understand the comparative effectiveness of buprenorphine vs. methadone in pregnancy, the impact of patient problem severity and treatment program structure on maternal (vs. neonatal) outcomes must be compared.

Significance:

Findings from this project will provide the preliminary data to support a comparative effectiveness clinical trial designed to compare the impact of office-based buprenorphine vs. federally licensed methadone programs on maternal treatment and postpartum functional outcomes in OD women. The ultimate goal of this line of research is develop evidence-based clinical guidelines to guide provider decision-making regarding the most effective treatment (buprenorphine vs. methadone) for a particular patient during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18+ years old, with a singleton pregnancy ≤ 28 weeks gestation confirmed by ultrasound, who meet Diagnostic and Statistical Manual-IV criteria for opioid dependence confirmed by urine drug screen (UDS), who are interested in opioid maintenance treatment and plan to receive prenatal care and deliver at Magee Womens Hospital (MWH) will be recruited.

Exclusion Criteria:

* (1) active, current dependence on benzodiazepines or alcohol
* (2) acute severe psychiatric condition in need of immediate treatment (e.g. suicidal ideations)
* (3) pending or legal action that could prohibit or interfere with participation (e.g. incarceration)
* (4) current, established treatment with methadone or buprenorphine. Exclusion criteria are based on the Substance Abuse and Mental Health Services Administration (SAMHSA) recommendations for office-based buprenorphine use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Number of participants who are recruited, enrolled, retained, and who complete the study. | 12 Months
  evaluate a minimum of 9 OD pregnant women per month for possible participation and enrollment, randomize a minimum of 4 participants per month to office-based buprenorphine (PRC) or methadone treatment facility (NATP) for a total of 50 participants over a 12 month enrollment period, retain ≥ 80% of randomized participants until 12 weeks postpartum, and maintain < 5% of incomplete data.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Krans, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Background] Meyer MC, Johnston AM, Crocker AM, Heil SH. Methadone and buprenorphine for opioid dependence during pregnancy: a retrospective cohort study. J Addict Med. 2015 Mar-Apr;9(2):81-6. doi: 10.1097/ADM.0000000000000092. PMID 25622120
- [Background] Jones HE, Heil SH, Baewert A, Arria AM, Kaltenbach K, Martin PR, Coyle MG, Selby P, Stine SM, Fischer G. Buprenorphine treatment of opioid-dependent pregnant women: a comprehensive review. Addiction. 2012 Nov;107 Suppl 1(0 1):5-27. doi: 10.1111/j.1360-0443.2012.04035.x. PMID 23106923
- [Background] Goodman D. Buprenorphine for the treatment of perinatal opioid dependence: pharmacology and implications for antepartum, intrapartum, and postpartum care. J Midwifery Womens Health. 2011 May-Jun;56(3):240-7. doi: 10.1111/j.1542-2011.2011.00049.x. PMID 21535372
- [Background] Fischer G, Gombas W, Eder H, Jagsch R, Peternell A, Stuhlinger G, Pezawas L, Aschauer HN, Kasper S. Buprenorphine versus methadone maintenance for the treatment of opioid dependence. Addiction. 1999 Sep;94(9):1337-47. doi: 10.1046/j.1360-0443.1999.94913376.x. PMID 10615719
- [Background] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR, Fischer G. Neonatal abstinence syndrome after methadone or buprenorphine exposure. N Engl J Med. 2010 Dec 9;363(24):2320-31. doi: 10.1056/NEJMoa1005359. PMID 21142534
- [Background] Jones ES, Fiellin DA. Women and opioid dependence treatment: office-based versus opioid treatment program-based care? Subst Abus. 2007 Jun;28(2):3-8. doi: 10.1300/J465v28n02_02. PMID 19266708
- [Background] Korthuis PT, Gregg J, Rogers WE, McCarty D, Nicolaidis C, Boverman J. Patients' Reasons for Choosing Office-based Buprenorphine: Preference for Patient-Centered Care. J Addict Med. 2010 Dec;4(4):204-10. doi: 10.1097/ADM.0b013e3181cc9610. PMID 21170143
- [Background] Hansen HB, Siegel CE, Case BG, Bertollo DN, DiRocco D, Galanter M. Variation in use of buprenorphine and methadone treatment by racial, ethnic, and income characteristics of residential social areas in New York City. J Behav Health Serv Res. 2013 Jul;40(3):367-77. doi: 10.1007/s11414-013-9341-3. PMID 23702611
- [Background] Moore BA, Fiellin DA, Barry DT, Sullivan LE, Chawarski MC, O'Connor PG, Schottenfeld RS. Primary care office-based buprenorphine treatment: comparison of heroin and prescription opioid dependent patients. J Gen Intern Med. 2007 Apr;22(4):527-30. doi: 10.1007/s11606-007-0129-0. PMID 17372805
- [Background] Fiellin DA, Schottenfeld RS, Cutter CJ, Moore BA, Barry DT, O'Connor PG. Primary care-based buprenorphine taper vs maintenance therapy for prescription opioid dependence: a randomized clinical trial. JAMA Intern Med. 2014 Dec;174(12):1947-54. doi: 10.1001/jamainternmed.2014.5302. PMID 25330017
- [Background] Jones ES, Moore BA, Sindelar JL, O'Connor PG, Schottenfeld RS, Fiellin DA. Cost analysis of clinic and office-based treatment of opioid dependence: results with methadone and buprenorphine in clinically stable patients. Drug Alcohol Depend. 2009 Jan 1;99(1-3):132-40. doi: 10.1016/j.drugalcdep.2008.07.013. Epub 2008 Sep 19. PMID 18804923
- [Background] Fiellin DA, Kleber H, Trumble-Hejduk JG, McLellan AT, Kosten TR. Consensus statement on office-based treatment of opioid dependence using buprenorphine. J Subst Abuse Treat. 2004 Sep;27(2):153-9. doi: 10.1016/j.jsat.2004.06.005. PMID 15450648
- [Background] Stine SM, Heil SH, Kaltenbach K, Martin PR, Coyle MG, Fischer G, Arria AM, Selby P, Jones HE. Characteristics of opioid-using pregnant women who accept or refuse participation in a clinical trial: screening results from the MOTHER study. Am J Drug Alcohol Abuse. 2009;35(6):429-33. doi: 10.3109/00952990903374080. PMID 20014912
- [Background] Almario CV, Seligman NS, Dysart KC, Berghella V, Baxter JK. Risk factors for preterm birth among opiate-addicted gravid women in a methadone treatment program. Am J Obstet Gynecol. 2009 Sep;201(3):326.e1-6. doi: 10.1016/j.ajog.2009.05.052. Epub 2009 Jul 24. PMID 19631928
- [Background] Cleary BJ, Donnelly JM, Strawbridge JD, Gallagher PJ, Fahey T, White MJ, Murphy DJ. Methadone and perinatal outcomes: a retrospective cohort study. Am J Obstet Gynecol. 2011 Feb;204(2):139.e1-9. doi: 10.1016/j.ajog.2010.10.004. Epub 2010 Dec 8. PMID 21145035
- [Background] Fischer G, Ortner R, Rohrmeister K, Jagsch R, Baewert A, Langer M, Aschauer H. Methadone versus buprenorphine in pregnant addicts: a double-blind, double-dummy comparison study. Addiction. 2006 Feb;101(2):275-81. doi: 10.1111/j.1360-0443.2006.01321.x. PMID 16445556
- [Background] Lacroix I, Berrebi A, Garipuy D, Schmitt L, Hammou Y, Chaumerliac C, Lapeyre-Mestre M, Montastruc JL, Damase-Michel C. Buprenorphine versus methadone in pregnant opioid-dependent women: a prospective multicenter study. Eur J Clin Pharmacol. 2011 Oct;67(10):1053-9. doi: 10.1007/s00228-011-1049-9. Epub 2011 May 3. PMID 21538146
- [Background] Mattick RP, Kimber J, Breen C, Davoli M. Buprenorphine maintenance versus placebo or methadone maintenance for opioid dependence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD002207. doi: 10.1002/14651858.CD002207.pub3. PMID 18425880
- [Background] Whitley SD, Sohler NL, Kunins HV, Giovanniello A, Li X, Sacajiu G, Cunningham CO. Factors associated with complicated buprenorphine inductions. J Subst Abuse Treat. 2010 Jul;39(1):51-7. doi: 10.1016/j.jsat.2010.04.001. PMID 20682186
- [Background] Teruya C, Schwartz RP, Mitchell SG, Hasson AL, Thomas C, Buoncristiani SH, Hser YI, Wiest K, Cohen AJ, Glick N, Jacobs P, McLaughlin P, Ling W. Patient perspectives on buprenorphine/naloxone: a qualitative study of retention during the starting treatment with agonist replacement therapies (START) study. J Psychoactive Drugs. 2014 Nov-Dec;46(5):412-26. doi: 10.1080/02791072.2014.921743. PMID 25364994
- [Background] Potter JS, Marino EN, Hillhouse MP, Nielsen S, Wiest K, Canamar CP, Martin JA, Ang A, Baker R, Saxon AJ, Ling W. Buprenorphine/naloxone and methadone maintenance treatment outcomes for opioid analgesic, heroin, and combined users: findings from starting treatment with agonist replacement therapies (START). J Stud Alcohol Drugs. 2013 Jul;74(4):605-13. doi: 10.15288/jsad.2013.74.605. PMID 23739025
- [Background] Jones HE, Johnson RE, Jasinski DR, O'Grady KE, Chisholm CA, Choo RE, Crocetti M, Dudas R, Harrow C, Huestis MA, Jansson LM, Lantz M, Lester BM, Milio L. Buprenorphine versus methadone in the treatment of pregnant opioid-dependent patients: effects on the neonatal abstinence syndrome. Drug Alcohol Depend. 2005 Jul;79(1):1-10. doi: 10.1016/j.drugalcdep.2004.11.013. PMID 15943939
- [Background] Holbrook AM, Jones HE, Heil SH, Martin PR, Stine SM, Fischer G, Coyle MG, Kaltenbach K. Induction of pregnant women onto opioid-agonist maintenance medication: an analysis of withdrawal symptoms and study retention. Drug Alcohol Depend. 2013 Sep 1;132(1-2):329-34. doi: 10.1016/j.drugalcdep.2013.02.031. Epub 2013 Mar 21. PMID 23523131
- [Background] Fiellin DA. The first three years of buprenorphine in the United States: experience to date and future directions. J Addict Med. 2007 Jun;1(2):62-7. doi: 10.1097/ADM.0b013e3180473c11. PMID 21768936
- [Background] Barry DT, Irwin KS, Jones ES, Becker WC, Tetrault JM, Sullivan LE, Hansen H, O'Connor PG, Schottenfeld RS, Fiellin DA. Integrating buprenorphine treatment into office-based practice: a qualitative study. J Gen Intern Med. 2009 Feb;24(2):218-25. doi: 10.1007/s11606-008-0881-9. Epub 2008 Dec 17. PMID 19089500
- [Background] Benoit E, Young R, Magura S, Staines GL. The impact of welfare reform on methadone treatment: policy lessons from service providers in New York city. Subst Use Misuse. 2004;39(13-14):2355-90. doi: 10.1081/ja-200034643. PMID 15603008
- [Background] Morgenstern J, Hogue A, Dauber S, Dasaro C, McKay JR. A practical clinical trial of coordinated care management to treat substance use disorders among public assistance beneficiaries. J Consult Clin Psychol. 2009 Apr;77(2):257-69. doi: 10.1037/a0014489. PMID 19309185
- [Background] Nunn A, Zaller N, Dickman S, Trimbur C, Nijhawan A, Rich JD. Methadone and buprenorphine prescribing and referral practices in US prison systems: results from a nationwide survey. Drug Alcohol Depend. 2009 Nov 1;105(1-2):83-8. doi: 10.1016/j.drugalcdep.2009.06.015. Epub 2009 Jul 21. PMID 19625142
- [Background] Roman PM, Abraham AJ, Rothrauff TC, Knudsen HK. A longitudinal study of organizational formation, innovation adoption, and dissemination activities within the National Drug Abuse Treatment Clinical Trials Network. J Subst Abuse Treat. 2010 Jun;38 Suppl 1:S44-52. doi: 10.1016/j.jsat.2009.12.008. PMID 20307795
- [Background] Simpson DD. A conceptual framework for drug treatment process and outcomes. J Subst Abuse Treat. 2004 Sep;27(2):99-121. doi: 10.1016/j.jsat.2004.06.001. PMID 15450644
- [Background] Andersen R, Chen MS, Aday LA, Cornelius L. Health status and medical care utilization. Health Aff (Millwood). 1987 Spring;6(1):136-56. doi: 10.1377/hlthaff.6.1.136. No abstract available. PMID 3583214
- [Background] Binder T, Vavrinkova B. Prospective randomised comparative study of the effect of buprenorphine, methadone and heroin on the course of pregnancy, birthweight of newborns, early postpartum adaptation and course of the neonatal abstinence syndrome (NAS) in women followed up in the outpatient department. Neuro Endocrinol Lett. 2008 Feb;29(1):80-6. PMID 18283247
- [Background] Winhusen T, Wilder C, Wexelblatt SL, Theobald J, Hall ES, Lewis D, Van Hook J, Marcotte M. Design considerations for point-of-care clinical trials comparing methadone and buprenorphine treatment for opioid dependence in pregnancy and for neonatal abstinence syndrome. Contemp Clin Trials. 2014 Sep;39(1):158-65. doi: 10.1016/j.cct.2014.08.009. Epub 2014 Aug 23. PMID 25183042
- [Background] Deverka PA, Lavallee DC, Desai PJ, Esmail LC, Ramsey SD, Veenstra DL, Tunis SR. Stakeholder participation in comparative effectiveness research: defining a framework for effective engagement. J Comp Eff Res. 2012 Mar;1(2):181-194. doi: 10.2217/cer.12.7. PMID 22707880
- [Background] Krans EE, Davis MM. Preventing Low Birthweight: 25 years, prenatal risk, and the failure to reinvent prenatal care. Am J Obstet Gynecol. 2012 May;206(5):398-403. doi: 10.1016/j.ajog.2011.06.082. Epub 2011 Jun 29. PMID 21889122
- [Background] Krans EE, Davis MM, Palladino CL. Disparate patterns of prenatal care utilization stratified by medical and psychosocial risk. Matern Child Health J. 2013 May;17(4):639-45. doi: 10.1007/s10995-012-1040-9. PMID 22581379
- [Background] Krans EE, Davis MM, Schwarz EB. Psychosocial risk, prenatal counseling and maternal behavior: findings from PRAMS, 2004-2008. Am J Obstet Gynecol. 2013 Feb;208(2):141.e1-7. doi: 10.1016/j.ajog.2012.11.017. Epub 2012 Nov 15. PMID 23159699
- [Background] Krans EE, Moloci NM, Housey MT, Davis MM. Impact of psychosocial risk factors on prenatal care delivery: a national provider survey. Matern Child Health J. 2014 Dec;18(10):2362-70. doi: 10.1007/s10995-014-1476-1. PMID 24740719
- [Background] McLellan AT, Kushner H, Metzger D, Peters R, Smith I, Grissom G, Pettinati H, Argeriou M. The Fifth Edition of the Addiction Severity Index. J Subst Abuse Treat. 1992;9(3):199-213. doi: 10.1016/0740-5472(92)90062-s. PMID 1334156
- [Background] Etter JF. A comparison of the content-, construct- and predictive validity of the cigarette dependence scale and the Fagerstrom test for nicotine dependence. Drug Alcohol Depend. 2005 Mar 7;77(3):259-68. doi: 10.1016/j.drugalcdep.2004.08.015. PMID 15734226
- [Background] Madden JD, Chappel JN, Zuspan F, Gumpel J, Mejia A, Davis R. Observation and treatment of neonatal narcotic withdrawal. Am J Obstet Gynecol. 1977 Jan 15;127(2):199-201. doi: 10.1016/s0002-9378(16)33250-1. PMID 831502
- [Background] Burns L, Conroy E, Mattick RP. Infant mortality among women on a methadone program during pregnancy. Drug Alcohol Rev. 2010 Sep;29(5):551-6. doi: 10.1111/j.1465-3362.2010.00176.x. PMID 20887580
- [Background] Bandstra ES, Morrow CE, Mansoor E, Accornero VH. Prenatal drug exposure: infant and toddler outcomes. J Addict Dis. 2010 Apr;29(2):245-58. doi: 10.1080/10550881003684871. PMID 20407980
- [Background] Creanga AA, Sabel JC, Ko JY, Wasserman CR, Shapiro-Mendoza CK, Taylor P, Barfield W, Cawthon L, Paulozzi LJ. Maternal drug use and its effect on neonates: a population-based study in Washington State. Obstet Gynecol. 2012 May;119(5):924-33. doi: 10.1097/AOG.0b013e31824ea276. PMID 22525903
- [Background] Jones HE, Heil SH, O'Grady KE, Martin PR, Kaltenbach K, Coyle MG, Stine SM, Selby P, Arria AM, Fischer G. Smoking in pregnant women screened for an opioid agonist medication study compared to related pregnant and non-pregnant patient samples. Am J Drug Alcohol Abuse. 2009;35(5):375-80. doi: 10.1080/00952990903125235. PMID 20180667
- [Background] Keegan J, Parva M, Finnegan M, Gerson A, Belden M. Addiction in pregnancy. J Addict Dis. 2010 Apr;29(2):175-91. doi: 10.1080/10550881003684723. PMID 20407975
- [Background] Chisolm MS, Tuten M, Brigham EC, Strain EC, Jones HE. Relationship between cigarette use and mood/anxiety disorders among pregnant methadone-maintained patients. Am J Addict. 2009 Sep-Oct;18(5):422-9. doi: 10.3109/10550490903077721. PMID 19874163
- [Background] Feske U, Tarter RE, Kirisci L, Pilkonis PA. Borderline personality and substance use in women. Am J Addict. 2006 Mar-Apr;15(2):131-7. doi: 10.1080/10550490500528357. PMID 16595350
- [Background] Peles E, Schreiber S, Naumovsky Y, Adelson M. Depression in methadone maintenance treatment patients: rate and risk factors. J Affect Disord. 2007 Apr;99(1-3):213-20. doi: 10.1016/j.jad.2006.09.017. Epub 2006 Oct 19. PMID 17055063
- [Background] Tuten M, Heil SH, O'Grady KE, Fitzsimons H, Chisolm MS, Jones HE. The impact of mood disorders on the delivery and neonatal outcomes of methadone-maintained pregnant patients. Am J Drug Alcohol Abuse. 2009;35(5):358-63. doi: 10.1080/00952990903108231. PMID 20180664
- [Background] Benningfield MM, Arria AM, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Fischer G, Jones HE, Martin PR. Co-occurring psychiatric symptoms are associated with increased psychological, social, and medical impairment in opioid dependent pregnant women. Am J Addict. 2010 Sep-Oct;19(5):416-21. doi: 10.1111/j.1521-0391.2010.00064.x. PMID 20716304
- [Background] Chatham LR, Hiller ML, Rowan-Szal GA, Joe GW, Simpson DD. Gender differences at admission and follow-up in a sample of methadone maintenance clients. Subst Use Misuse. 1999 Jun;34(8):1137-65. doi: 10.3109/10826089909039401. PMID 10359226
- [Background] Ashley OS, Marsden ME, Brady TM. Effectiveness of substance abuse treatment programming for women: a review. Am J Drug Alcohol Abuse. 2003;29(1):19-53. doi: 10.1081/ada-120018838. PMID 12731680
- [Background] Rowan-Szal GA, Chatham LR, Joe GW, Simpson DD. Services provided during methadone treatment. A gender comparison. J Subst Abuse Treat. 2000 Jul;19(1):7-14. doi: 10.1016/s0740-5472(99)00091-4. PMID 10867295
- [Background] Latt NC, Spencer JD, Beeby PJ, McCaughan GW, Saunders JB, Collins E, Cossart YE. Hepatitis C in injecting drug-using women during and after pregnancy. J Gastroenterol Hepatol. 2000 Feb;15(2):175-81. doi: 10.1046/j.1440-1746.2000.02060.x. PMID 10735542
- [Background] Dashe JS, Jackson GL, Olscher DA, Zane EH, Wendel GD Jr. Opioid detoxification in pregnancy. Obstet Gynecol. 1998 Nov;92(5):854-8. doi: 10.1016/s0029-7844(98)00312-3. PMID 9794682
- [Background] Stewart RD, Nelson DB, Adhikari EH, McIntire DD, Roberts SW, Dashe JS, Sheffield JS. The obstetrical and neonatal impact of maternal opioid detoxification in pregnancy. Am J Obstet Gynecol. 2013 Sep;209(3):267.e1-5. doi: 10.1016/j.ajog.2013.05.026. Epub 2013 May 29. PMID 23727040
- [Background] Jones HE, Finnegan LP, Kaltenbach K. Methadone and buprenorphine for the management of opioid dependence in pregnancy. Drugs. 2012 Apr 16;72(6):747-57. doi: 10.2165/11632820-000000000-00000. PMID 22512363
- [Background] Jones HE, Deppen K, Hudak ML, Leffert L, McClelland C, Sahin L, Starer J, Terplan M, Thorp JM Jr, Walsh J, Creanga AA. Clinical care for opioid-using pregnant and postpartum women: the role of obstetric providers. Am J Obstet Gynecol. 2014 Apr;210(4):302-310. doi: 10.1016/j.ajog.2013.10.010. Epub 2013 Oct 10. PMID 24120973
- [Background] Krans EE, Cochran G, Bogen DL. Caring for Opioid-dependent Pregnant Women: Prenatal and Postpartum Care Considerations. Clin Obstet Gynecol. 2015 Jun;58(2):370-9. doi: 10.1097/GRF.0000000000000098. PMID 25775440